CLINICAL TRIAL: NCT06968923
Title: Effectiveness of a Home-Based Rehabilitation Program in Stroke Survivors Using the Euleria Home® Device: A Crossover Study.
Brief Title: Effectiveness of a Home-Based Rehabilitation Program in Stroke Survivors Using the Euleria Home® Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Professor, Universita di Verona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1742CESC
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Telemedicine; Rehabilitation; Telerehabilitation
Keywords: Stroke; telemedicine; telerehabilitation; motor; cognitive
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): The group undergoes a 5-week treatment, twice a week, for a total of 10 rehabilitation sessions. Each session lasts approximately 60 minutes. The treatment follows standard in-person clinical practice.
- Group B (Experimental): The group undergoes a 5-week treatment, with 2 hours per week, for a total of 10 hours at home. Each session lasts approximately 20 minutes. The treatment consists of a sequence of exercises performed using the Euleria Home® device, a medical software that enables the delivery of personalized exercise therapy programs designed by a healthcare professional.
  Interventions: Behavioral: Telerehabilitation

INTERVENTIONS:
Behavioral: in person treatment — The group undergoes a 5-week treatment, twice a week, for a total of 10 rehabilitation sessions. Each session lasts approximately 60 minutes. The treatment follows standard in-person clinical practice.
Behavioral: Telerehabilitation — The group undergoes a 5-week treatment, with 2 hours per week, for a total of 10 hours at home. Each session lasts approximately 20 minutes. The treatment consists of a sequence of exercises performed using the Euleria Home® device, a medical software that enables the delivery of personalized exercise therapy programs designed by a healthcare professional.
  Arms: Group B

SUMMARY:
To verify the non-inferiority, in terms of post-treatment (T1) clinical effectiveness, of a "multidomain" telerehabilitation (TR) protocol compared to conventional outpatient rehabilitation in patients with stroke sequelae, with respect to motor, cognitive, and language functions. The absence of statistically significant differences between the two groups regarding treatment effects for each targeted domain will be considered an indicator of non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* First diagnosis of ischemic stroke, documented radiologically via CT or MRI scans, corresponding to ICD-9-CM codes 433 and 434 .
* Presence of aphasia, as assessed by the Aachener Aphasia Test (AAT), and/or cognitive deficits identified through the Oxford Cognitive Screen (OCS).
* Availability of an ADSL or higher-speed internet connection at the patient's residence.
* Ability of the patient and/or caregiver to understand and utilize the telerehabilitation system.
* Provision of written informed consent.

Exclusion Criteria:

* Contemporanea partecipazione ad altri studi clinici;
* Decadimento cognitivo
* Deformità ossee come conseguenza di precedenti eventi traumatici ai 4 arti;
* Contratture fisse ai 4 arti valutate come 4/4 alla scala di Ashworth modificata (MAS)
* Altre patologie neurologiche e ortopediche in grado di interferire con lo studio.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper and Lower Limb (FMA) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  The Fugl-Meyer Assessment (FMA) is a widely used observational scale for evaluating motor recovery in patients with stroke sequelae. In its version focused on the upper and lower limbs, the FMA measures motor control by assessing specific movements of the shoulder, elbow, wrist, hand, hip, knee, and ankle. Each movement is rated on a three-point scale (0 = absent, 1 = partial, 2 = complete). The maximum score is 66 points for the upper limb and 34 for the lower limb, for a total of 100 points in the overall motor function assessment. Higher scores indicate a greater degree of recovery.

SECONDARY OUTCOMES:
The Trail Making Test - A (TMT-A) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  Used as a measure of psychomotor speed and visual search/attention skills
Trail Making Test Part B (TMT-B) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  Used as a measure of attentional set-shifting and mental flexibility. Time needed to complete the tasks is recorded.
Berg Balance Scale (BBS) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A clinical assessment of balance that assigns an overall score ranging from 0 to 56, where a higher score indicates good balance control and a reduced risk of falls.
10 Meters Walking Test (10MWT) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  An assessment that measures a person's walking speed over a distance of 10 meters. During the test, the patient walks at a comfortable pace, and the time taken to cover the 10 meters is recorded.
Timed Up and Go (TUG) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A test to measure a person's level of mobility, requiring both static and dynamic balance skills. It measures the time it takes for a person to stand up from a chair, walk three meters, turn around, return to the chair, and sit down again.
Barthel Index (BI) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A scale used to assess a person's autonomy in daily activities, such as eating, dressing, walking, and other motor and self-care functions. Composed of 10 items, the score ranges from 0 to 100, with higher scores indicating greater independence in daily activities, while lower scores reflect greater dependence or the need for assistance.
Short Form - 36 (SF-36) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A questionnaire used to assess changes in a person's health status, considering various dimensions of physical and mental well-being. Composed of 36 questions, the SF-36 explores areas such as physical health, pain, the ability to perform daily activities, vitality, emotional health, social functioning, and mental health.
Client Satisfaction Questionnaire (CSQ-8) | The test is administered after five weeks of treatment, and four weeks post-treatment.
  a self-administered post-treatment questionnaire, comprised of eight items that evaluate the level of satisfaction regarding the care and quality of the service received and the level of fulfillment of the patient's expectations regarding the treatment administered. The total score of the questionnaire is 32 points, with higher values meaning higher satisfaction with the treatment received.
Oxford Cognitive Screen (OCS) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A neuropsychological assessment tool that measures a person's global cognitive status, providing an analysis of key cognitive functions such as memory, executive functions, praxis, attention, language, and visuospatial exploration. Composed of various sub-tests, the OCS allows for the rapid and systematic identification of potential cognitive deficits and is particularly useful in patients with brain damage, such as those with stroke.
Digit Span Forward (DSF) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A test that measures short-term memory, specifically the ability to retain and recall sequences of numbers. During the test, the patient is asked to repeat a series of numbers read aloud by the examiner, starting with a short sequence and progressively increasing the length. The patient's performance is assessed based on the maximum number of digits they can correctly repeat in the same order as presented.
Digit Span Backward | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A test that evaluates working memory, a cognitive function that allows the temporary storage and manipulation of information. In this test, the patient is asked to repeat a sequence of numbers read by the examiner, but in reverse order from how they were presented. The difficulty progressively increases with the addition of more digits in the sequence.
Frontal Assessment Battery (FABit) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  A neuropsychological test that evaluates basic executive functions, including abilities such as abstraction, verbal ideation, sensitivity to interference, motor planning, inhibitory control, and environmental dependence. It has a maximum total score of 18 points, divided into 6 sub-tests, each of which can assign up to 3 points. High scores indicate preserved executive functioning.
Symbol Digit Modalities Test | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  This test evaluates the visual information processing speed and attention; the number of correct answers in 90 seconds is registered (higher scores indicate better performance).
Hospital Anxiety and Depression Scale (HADS) | The test is administered at the beginning of the treatment (> six months after the event), after five weeks of treatment, and four weeks post-treatment.
  HADS is a self-report questionnaire commonly used to assess emotional distress in medical patients, specifically focusing on symptoms of anxiety and depression. It consists of 14 items, with 7 items dedicated to anxiety (HADS-A) and 7 to depression (HADS-D). Each item is rated on a 4-point Likert scale ranging from 0 to 3, reflecting the intensity or frequency of symptoms over the past week. The maximum score is 21 for each subscale, with higher scores indicating greater symptom severity. Scores from 0 to 7 are considered within the normal range, 8 to 10 suggest borderline abnormal levels, and 11 or above indicate clinically significant anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona - UOC di Neuroriabilitazione, Verona, verona, Italy